CLINICAL TRIAL: NCT05610098
Title: Comparing Gene Expression Profiles of Adults With Isolated Spinal TB to Disseminated Spinal TB Identified by 18FDG-PET/CT at Time of Diagnosis, 6-and 12-months Follow-up
Brief Title: Gene Expression Profiles in Spinal Tuberculosis.
Acronym: SpinalTBX
Status: Recruiting | Type: Observational
Sponsor: University of Cape Town (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Prof Friedrich Thienemann, Professor, Principal Investigator and Research Group Leader, University of Cape Town
Other Study IDs: HREC 243/2022; AOS-DIA-22-029-TRA (Other Grant/Funding Number: AO Foundation)
Record Dates: First submitted 2022-10-24; First posted 2022-11-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis, Spinal; Tuberculosis, Osteoarticular; Tuberculosis; Mycobacterium Infections; Infections; Bone Diseases, Infectious; Musculoskeletal Diseases; Spinal Disease; Spondylitis; Spondylitis; Tuberculosis (Manifestation); Spondylodiscitis; Positron-Emission Tomography; Diagnostic Imaging; Diagnostic Techniques and Procedures
Keywords: Spinal TB; tuberculous spondylodiscitis; FDG-PET/CT; POC
MeSH Terms: conditions — Tuberculosis, Spinal; Tuberculosis, Osteoarticular; Tuberculosis; Mycobacterium Infections; Infections; Bone Diseases, Infectious; Musculoskeletal Diseases; Spinal Diseases; Spondylitis; Discitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Site of disease specimen collection (sputum, spinal abscess/disc/bone tissue collection); whole-blood samples, serum, PBMC, Paxgene.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tuberculosis (TB) is one of the top ten causes of death worldwide with approximately 10 million cases globally and 1.2 million deaths. Sub-Saharan Africa carries the highest burden of TB. South Africa has one of the highest HIV and TB rates worldwide with an HIV prevalence rate in adults of 19% and a TB case notification rate of 615/100,000 in 2019. Over many years, focus has been paid to pulmonary TB and extrapulmonary TB (EPTB) has received only little attention even though it accounts for almost a quatre of all TB cases. The diagnosis of EPTB remains challenging simply because sample collection requires invasive procedures in the absence of a blood-based diagnostic test. Spinal TB (spondylitis or spondylodiscitis caused by Mycobacterium tuberculosis) - often known as Pott's disease - accounts for up to 10% of EPTB and affects young children, people with HIV-coinfection and elderly, and often leads to lifelong debilitating disease due to devastating deformation of the spine and compression of neural structures. Little is known with regards to the extent of disease and isolated TB spine as well as a disseminated form of TB spine have been described. The latter presents with a spinal manifestation plus disseminations to other organs such as the lungs, pleura, lymph nodes, the GIT or urinary tract or even the brain.

In the Spinal TB X cohort, the investigators aim to describe the clinical phenotype of spinal TB using whole body PET/CT and identify a specific gene expression profile for the different stages of dissemination and compare findings to previously described signatures for latent and active pulmonary TB. A blood-based test for spinal TB would lead to earlier diagnosis and treatment in all settings globally and improve treatment outcome of this devastating disease.

DETAILED DESCRIPTION:
In the Spinal TB X cohort, the investigators aim to describe the clinical phenotype of spinal TB using whole body PET/CT and identify a specific gene expression profile for the different stages of dissemination and compare findings to previously described signatures for latent and active pulmonary TB. A blood-based test for spinal TB would lead to earlier diagnosis and treatment in all settings globally and improve treatment outcome of this devastating disease.

1. The investigators hypothesize that spinal TB may present as two clinical phenotypes: isolated spinal TB with no additional lesion on whole body PET/CT and disseminated spinal TB with a spinal lesion plus an additional extraspinal lesion on whole body PET/CT.
2. The investigators hypothesize that a specific gene expression profile may distinguish between the two clinical entities above and allows for treatment monitoring during antimicrobial therapy ("personalized medicine")
3. The investigators hypothesize that whole body PET/CT is superior to MRI in diagnosing spinal and extraspinal TB.

Primary objective

To describe the clinical phenotype of spinal TB using whole body PET/CT and to identify mRNA gene expression profiles of isolated spinal TB versus disseminated spinal TB stratified by HIV status.

Secondary objectives

1. To identify the distributive patterns of suspected spinal TB using two imaging modalities: MRI and PET/CT.
2. To analyse the genomes of Mtb. extracted from different sites of the body (if available) and to identify differences in their genome regarding SNPs and drug sensibility.
3. To analyse imaging findings using PET/CT at treatment initiation, 6 months, and 12 months to better understand treatment outcome using PET/CT.
4. To compare imaging findings on PET/CT and MRI at baseline to evaluate the role of PET/CT in spinal TB diagnostics (virtual biopsy).

Design

This is a prospective cohort study to develop new diagnostics for isolated spinal TB versus disseminated spinal TB and treatment monitoring. Furthermore, this study investigates genetic variability in spinal TB and its distributional pattern. After MRI-confirmation of spinal TB according to local algorithms, patients will be included in the study. At baseline, clinical examination as well as blood collection will be performed. Every patient with no confirmed HIV will undergo HIV-testing. Sputum will be collected and screening for diabetes and pregnancy will be completed. Whole-body PET/CTs will be performed at 0 months, 6 months, and 12 months. Spinal biopsies will be gathered if surgery is being performed. Samples of the sites of disease will be acquired if applicable and TB culture as well as GeneXpert will be performed.

Recruitment

Patients with newly diagnosed spinal TB at the Department of Orthopaedics, Groote Schuur Hospital, Cape Town, South Africa.

ELIGIBILITY:
Inclusion Criteria

1. Participant has completed the written informed consent process prior to undergoing any clinical evaluations and willing to undergo HIV testing
2. TB spine based on clinical and radiological criteria
3. Age 18 or older with a body weight of at least 40 kg body weight
4. Able and willing to return to follow-up
5. Willing to have samples, including DNA including RNA extraction, stored
6. Willing to consistently practice a highly reliable method of pregnancy prevention

Exclusion Criteria

1. Pregnancy or active desire to become pregnant within the next 6 months.
2. Uncontrolled diabetes (HbA1c ≥ 6.5% / random glucose concentration ≥11.1 mmol/l, fasting plasma glucose ≥ 7.0 mmol/l)
3. Alcohol and substance abuse which might interfere with medication adherence during the trial
4. Positive SARS-CoV-2 PCR in the past 4 weeks
5. Suspicion of malignancy on MRI or known malignancy
6. Suspicion of inflammatory disease and other rheumatological conditions
7. Any person for whom the physician feels this study is not appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with clinically and MR-suspected spinal TB will be recruited from the Department of Orthopaedics, Groote Schuur Hospital, Cape Town, South Africa. According to the current caseload, the investigators will be able to include 50-100 participants per year, aiming for 100 participants in total. In result, the investigators are aiming for 300 PET/CTs (100 initial, 100 at 6 months, 100 at 12 months) and 300 peripheral blood samples for gene expression analysis.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical phenotype of spinal TB | 3 years
  To describe the clinical phenotype of spinal TB using whole body PET/CT a semiquantitative approach will be used. Regions of interest (ROIs) will be identified with increased FDG uptake against background and total lesion glycolysis (TLG) of each ROI will be measured using MIM software
mRNA gene expression profiles of spinal TB | 3 years
  mRNA gene expression profiles of isolated spinal TB versus disseminated spinal TB described in outcome 1 will be measured and stratified by HIV status.

SECONDARY OUTCOMES:
MRI vs. PET/CT at the site of disease (spine level) | 3 years
  To identify the distributive patterns of suspected spinal TB using two imaging modalities: MRI and PET/CT. MRI is measure T1, T2 and diffusion weighted images. Regions of interest (ROIs) in the spine will be identified with increased FDG uptake against background and total lesion glycolysis (TLG) of each ROI will be measured using MIM software
Whole Genome Sequencing of Mtb. isolates | 3 years
  To analyse the genomes of Mtb. extracted from different sites of the body (if available) and to identify differences in their genome regarding SNPs and drug sensibility.
PET/CT changes over 12 months | 3 years
  Regions of interest (ROIs) in the spine will be identified with increased FDG uptake against background and total lesion glycolysis (TLG) of each ROI will be measured using MIM software at different timepoints: treatment initiation, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: friedrich Thienemann, MD, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scherer J, Mukasa SL, Wolmarans K, Guler R, Kotze T, Song T, Dunn R, Laubscher M, Pape HC, Held M, Thienemann F. Comparing gene expression profiles of adults with isolated spinal tuberculosis to disseminated spinal tuberculosis identified by 18FDG-PET/CT at time of diagnosis, 6- and 12-months follow-up: classifying clinical stages of spinal tuberculosis and monitoring treatment response (Spinal TB X cohort study). J Orthop Surg Res. 2024 Jun 25;19(1):376. doi: 10.1186/s13018-024-04840-7. PMID 38918806
- See also: General Medicine & Global Health research group at the University of Cape Town — http://www.gmgh.africa